



Site: St Mary's Hospital Patient Hospital Number:

Subject Identification Number for this trial:

## CONSENT FORM Phase 1

Version 1.2, Date 12/05/2016

**Title of Project:** 

The Step Home Trial: Utilising Physical Activity Data in the Acute Post-operative Setting

## Name of Researcher:

Ms Aliza Abeles
Department of Surgery and Cancer
10<sup>th</sup> Floor QEQM building
St Mary's Hospital
Praed Street
London W2 1NY United Kingdom

Email: a.abeles@imperial.ac.uk

| | | | Please initial box |
|---|---|---|---|
| 1. | I confirm that I have read and understand the information sheet dated 12/05/2016 version 2.2 for the above study and have had the opportunity to ask questions. | | |
| 2. | , , , | understand that my participation is voluntary and that I am free to withdraw at any time, vithout giving any reason, without my medical care or legal rights being affected. | |
| to i | 3. I understand that sections of any of my medical notes may be looked at by responsible individuals from Imperial College, the NHS Trust or from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to access my records that are relevant to this research. | | |
| | . I understand that if I was to lose capacity to consent during the study, although no further data would be collected, the data already collected may still be used in the study. | | |
| 5. | I agree to take part in the above | study. | |
| <br>Na | me of Participant | Date | Signature |
| Name of Person taking consent (if different from researcher) | | Date | Signature |
| <br>Re | searcher | Date | Signature |

(COPIES: 1 for participant, 1 for researcher, 1 for medical notes)